CLINICAL TRIAL: NCT05628870
Title: A Single-arm, Open-label, Multi-center Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HRS-1358 Monotherapy or Combination With Dalpiciclib Isethionate Tablets in Patients With Metastatic or Locally Advanced Breast Cancer.
Brief Title: A Trial of HRS-1358 Tablets in Metastatic or Local Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1358-I-101
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm study of HRS-1358
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1358 (Experimental): Daily oral dosages of HR-1358； Daily oral dosages of HR-1358 and Dalpiciclib Isethionate Tablets
  Interventions: Drug: HRS-1358

INTERVENTIONS:
Drug: HRS-1358 — HRS-1358 or combination with Dalpiciclib Isethionate Tablets will be administered daily orally in continuous dosing over 28-day cycles.

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets in patients with metastatic or locally advanced breast cancer in order to estimate the Dose-Limiting Toxicity (DLT), Maximum Tolerated Dose (MTD) and select the Recommended Phase 2 Dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosis of local advanced or metastatic breast cancer
2. Women must be postmenopausal, or pre-/peri-menopausal women must be on ovarian suppression
3. At least 1 line of endocrine therapy in the metastatic or advanced setting
4. ECOG performance status score: 0-1;
5. Adequate organ functions as defined
6. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study.

Exclusion Criteria:

1. the investigators judged that it was not suitable to endocrine therapy
2. patients with active brain metastasis (without medical control or with clinical symptoms),
3. History of clinically significant cardiovascular or cerebrovascular diseases
4. The subject has one of many factors affecting oral 、absorption, distribution, metabolism and excretion of drugs
5. Active autoimmune diseases, History of immunodeficiency, including positive HIV serum test result and other acquired or congenital immunodeficiency diseases, or history of organ transplantation
6. Have received other similar drugs in the past;
7. Known history of allergy to HRS-1358 ingredients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicities (DLTs) | up to 28 days
  Number of participants with dose-limiting toxicities (DLTs)
Maximum tolerated dose | up to 28 days
  The Maximum tolerated dose of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
RP2D | Change From Baseline at 28 days
  select the Recommended Phase 2 Dose (RP2D) of HRS-1358 or combination with Dalpiciclib Isethionate Tablets
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | up to 30 days after the last dose
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Cmax | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Tmax | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
AUC0-t | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Cmax,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Tmax,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Cmin,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
AUCss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Rac | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fourth treatment period
  PK parameters of multiple doses of HRS-1358 monotherapy or combination with Dalpiciclib Isethionate Tablets
Overall response rate (ORR) in participants | Up to approximately 1 year
Clinical benefit rate (CBR) in participants | Up to approximately 1 year
Duration of response (DOR) in participants | Up to approximately 1 year
Progression Free Survival (PFS) observed in participants | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided